CLINICAL TRIAL: NCT02177825
Title: Phase II Study of Imatinib Mesylate in Neurofibromatosis Type I Patients Aged 2 to 21 With Plexiform Neurofibromas
Brief Title: Study of Imatinib Mesylate in Neurofibromatosis Type I Patients Aged 2 to 21 With Plexiform Neurofibromas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual 5 patients out of 25 expected. Primary objectives could not be met without recruiting more patients.
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Dr Perreault, Neurologist, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLNEU SJ 01
Record Dates: First submitted 2014-06-25; First posted 2014-06-30 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Plexiform Neurofibromas
MeSH Terms: conditions — Neurofibroma, Plexiform | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imatinib Mesylate (Experimental): Imatinib Mesylate at 110 mg/m2 up to 440mg/m2 PO per day for twelve months taken in one morning dose (if dose is less than 200 mg/day) or two doses (morning and evening)
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — oral administration
  Other Names: Imatinib

SUMMARY:
This phase II trial will test the hypothesis that inhibition of c-kit signalling pathways in pediatric patients with Neurofibromatosis Type I(NF-1) and progressing plexiform neurofibroma will result in objective reduction and/or inhibition of plexiform neurofibromas progression.

This will be a Phase II study of imatinib mesylate given orally. Patients with stable or responding disease may receive the drug for a period not exceeding one year.

DETAILED DESCRIPTION:
Clinical objectives

1. Demonstrate the clinical benefit of imatinib in a pediatric patient population with progressing and metabolically active plexiform neurofibromas (NF)
2. Demonstrate the need or not to pursue treatment for more than a year in responders to imatinib

Biological studies objectives

1. Identify biological markers of plexiform neurofibroma progression and response to treatment
2. Identify biological markers of mast cell responses to imatinib, given that mast cells are required for tumorigenesis and are a target for imatinib

Imaging studies objectives

Using 18-Fluorodeoxyglucose-positron Emission Tomography (FDG PET/CT):

1. Identify imaging characteristics of progressing plexiform neurofibromas
2. Assess the role of F18-FDG PET/CT in comparison with CT/MRI to evaluate response to imatinib ¸

Pharmacological study

1. Evaluate trough plasma levels of imatinib and its active metabolite (NDMIL N-desmethyl imatinib) achieved in this pediatric population
2. Identify potential correlation between imatinib (and NDMI) trough levels achieved and clinical response

ELIGIBILITY:
Inclusion Criteria:

1. Age Greater than or equal to 2 years and up to 21 years of age at time of study enrolment
2. Diagnosis Patients with NF1 and an inoperable plexiform NFs that has the potential to cause significant morbidity.
3. Patients must have measurable disease by magnetic resonance imaging (MRI) and progressive plexiform neurofibroma(s) with or without clinical symptoms.

   * Patients must have a recent FDG-PET scan imaging study done in the last 3 months before being offered participation to the study
   * Surgery/Residual disease: Patients are only eligible if complete tumor resection is not feasible, or if a patient with a surgical option refuses surgery. Evidence of recurrent or progressive disease is NOT necessary. Patients must be at least 21 days from surgery, if performed, prior to receiving their first dose of study drug
4. Performance level Patients must have a Karnofsky of > 70% or Lansky of >50% and a life expectancy of > 6 months.
5. Previous use of imatinib is permitted if there was no progressive disease during treatment.
6. Prior therapy Patients must be at least 28 days without any treatment before enrolment in this study.
7. Patient is free of another primary malignancy except if the other primary malignancy neither currently clinically significant nor requiring active intervention.
8. Organ function requirement

   * Creatinine < 1.5 x upper limit of normal (ULN)
   * Total bilirubin < 1.5 x ULN and SGOT and SGPT < 2.5 x ULN
   * ANC > 1.5 x 109/L and Platelets > 100 x 109/L
9. Reproductive potential Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.

Exclusion Criteria:

1. Patient has received any other investigational agents within 28 days of first day of study drug dosing.
2. Patient with rapidly progressing disease may be enrolled before the 28 days period. In these cases, only the study chair can take this decision.
3. Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria.
4. Female patients who are pregnant or breast-feeding.
5. Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection)
6. Patient has a known brain metastasis. Non-specific central nervous system (CNS) changes on MRI/CT characteristic of NF1 are allowed, but not known CNS malignancies.
7. Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
8. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
9. Patient received chemotherapy within 4 weeks prior to study entry.
10. Patient previously received radiotherapy to greater than or equal to 25% of the bone marrow within 24 months.
11. Patient had a major surgery within 2 weeks prior to study entry.
12. Patient with any significant history of non-compliance to medical regimens.
13. Patients who have or anticipate receiving permanent (or semi-permanent) metallic structures attached to their body. (e.g., braces on teeth, body piercings), which their physicians believe will interfere with the MRI.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2014-06; Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Demonstrate the clinical benefit of imatinib in a pediatric patient population with progressing and metabolically active plexiform NFs | 12 months
  Time to tumor progression as assessed by volumetric MRI and FDG-PETScan analysis at baseline, after 3, 6, 9, and 12 months on therapy.

SECONDARY OUTCOMES:
Changes in NF1 biomarkers after treatment with imatinib | 12 months
  Patients on imatinib will have blood samples and urine taken at baseline and every 3 months until treatment completion or until disease progression. Mastocyte activation biomarkers will be monitored and evaluated as potential disease state indicators.

OTHER OUTCOMES:
Evaluate trough plasma levels of imatinib and its active metabolite (NDMIL N-desmethyl imatinib) achieved in this pediatric population | 12 months
  We will evaluate trough plasma levels of imatinib achieved in this patient population at 3, 6, 9 and 12 month and correlate it with response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Perreault, MD/FRCPC, Principal Investigator — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada